CLINICAL TRIAL: NCT05735730
Title: Diet, Lifestyle, Systemic Medication and Genetics: Can the Risk for AMD be Modulated?
Brief Title: Can the Risk for AMD be Modulated?
Acronym: AMD_LifeGene
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4C-2022-11
Record Dates: First submitted 2022-12-22; First posted 2023-02-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-05

CONDITIONS: Age-Related Macular Degeneration (ARMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidemiologic study (Other): This is an epidemiologic study. No arms are considered.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — The study intervention consists of a blood draw for genetic analysis.

SUMMARY:
The goal of this Cross-sectional, interventional study is to learn about whether different risk factors, as Mediterranean diet, lifestyle and concomitant medication can modulate the risk imprinted by genetics in Age-related macular degeneration (AMD). The main question it aims to answer is: How the genetic risk interacts with environmental and lifestyle factors, especially Mediterranean diet and chronic medication, in order to assess how this interplay protects or presents higher risk for the establishment or the progression of AMD.

Participants:

Vital Signs will be measured; Medical History, Demographics, Nutritional/lifestyle habits and Family History of AMD will be recorded; Ophthalmological Examination will be performed Genetic analysis will be performed.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the major cause of vision loss in people over 55 years in western countries. By 2040, AMD prevalence is estimated to reach 288 million. Age-related macular degeneration is a multifactorial disease, implying genetic and demographic/environmental risk factors. Several worldwide epidemiologic studies characterized AMD from an epidemiologic standpoint, identifying risk factors for the disease, such as age and smoking habits, the two most widely accepted, besides genetics. Most of these studies have evaluated the different risk factors from a single-way point of view, not assessing gene-lifestyle/nutrition/medication interplay. A few studies stepped forward on this matter by studying the difference between the genetic risk conferred by specific and associated single nucleotide polymorphisms (SNPs), alone or in combination with other risk factors. Our group conducted the Epidemiological Study of the Prevalence of AMD in Portugal (NCT01298674) and assessed the prevalence of AMD in two cohorts (from an inland population - Lousã, and a costal one - Mira), and subsequently assessed the AMD incidence in the coastal cohort (Mira), in the Five-year Incidence of Age-related Macular Degeneration in the Central Region of Portugal study - AMDIncidencePT (NCT02748824). AMD prevalence in Mira was inferior to that in Lousã, emphasizing that this population may have specific environmental, lifestyle or genetic characteristics. Differences in major allele frequencies were already identified in the coastal population in the AMD incidence study (NCT02748824) that might explain the previous findings in both prevalence and incidence in the Mira population, and it was found that rare variants conferred high risk of disease in this coastal cohort. Increasing the sample and analysis of another geographic population by focusing now on the incidence and genetic data from the inland population of Lousã will further contribute to the disease genetic knowledge in Europe, and by extension, will deepen the knowledge on genetic interplay with environment and lifestyle, under the concept of personalized medicine. Therefore, data obtained in this study regarding the inland population cohort (Lousã) will also be analyzed together and compared with the data relative to the coastal population cohort (Mira) from the AMD incidence study (NCT02748824) and the Life Style and Food Habits Questionnaire in the Portuguese Population Aged 55 or More (NCT01715870).

The aim of the AMD_LifeGene study is to further explore the interplay between AMD risk factors and AMD genetic risk and their impact on AMD development. This study will allow the investigation of whether different risk factors, as the Mediterranean diet, lifestyle and concomitant medication can modulate the risk imprinted by genetics.

AMD_LifeGene is a cross-sectional, interventional study with no investigative treatment or medical device and with a single visit. The study intervention consists of a blood draw (for genetic and molecular analysis), that is not considered part of AMD routine care, for the participants that give consent for this procedure. Therefore, this is considered an interventional study in accordance with the Portuguese Clinical Research National Law 21/2014 of 16 of April amended by Law 73/2015 of 27 of July and Law 49/2018 of 14 August. The residents of the Lousã region who have already participated in the first study to determine the prevalence of AMD (NCT01298674), will be contacted to participate in the AMD_LifeGene study. Data collection will be carried out by AIBILI-CEC at the Lousã Healthcare Unit.

This study will have as primary endpoints: assessment of risk factors including demographics, medical history, ophthalmic history, family history of AMD, systemic co-morbidities and medication, nutritional/diet and lifestyle habits, together with a complete phenotypic characterization of AMD on multimodal imaging evaluation, and association with the genetic background. Secondary endpoints will be epidemiological characterization of this larger population that includes both the inland and coastal cohorts in terms of incidence and disease progression.

After signing the Informed Consent Form, participants will be submitted to a single visit approximately ten years after the participant's participation in the Epidemiological Study (NCT01298674). Data on participants' demographics, vital signs, medical history (general and ophthalmic), analytical systemic parameters, family history of AMD, current medication, and nutritional/diet and lifestyle habits will be collected. For those who give consent, a blood sample will be collected for molecular and genetic analysis.

Ophthalmologic examination will be performed on both eyes including visual acuity, tonometry, and multimodal imaging with Colour Fundus Photography (CFP), Spectral-Domain Optical Coherence Tomography (SD-OCT), OCT Angiography (OCTA), Fundus Autofluorescence (FAF), Infrared imaging (IR) and Ultra-Widefield Fundus Imaging (UWF-FI) / FAF.

Ophthalmological examinations performed will be analyzed at AIBILI Coimbra Ophthalmology Reading Centre (AIBILI-CORC).

All imaging data collected will be exported to AIBILI's Reading Centre (CORC) for centralized reading and grading, performed according to pre-specified grading protocols by certified ophthalmologist graders. The grading will be performed in two steps:

1. General grading: disease/no disease staging.
2. AMD phenotypic and stage grading: this assessment will be applicable to those eyes that were graded as AMD in the previous step.

Grading will be carried out by classifying the signs of AMD into 5 exclusive stages (stage 0-4) using the Rotterdam staging system, and additionally, with the Beckman classification system. The grading will be performed for both eyes. However, AMD staging, for an individual participant, will be based on the eye that presents a more severe status, if both eyes are gradable. If only one eye is gradable, the grading will be based only on it.

Genetic analysis will be performed by the International Age-Related Macular Degeneration Genomics Consortium (IAMDGC).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects residing in the Lousã region who participated in the epidemiologic study;
* Subjects capable of understanding the information about the study and to give their written informed consent to enter the study;
* Subjects willing and able to comply with the study procedures.

Exclusion Criteria:

- No exclusion criteria apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2028-01-12 (Estimated)

PRIMARY OUTCOMES:
Development of AMD | 18 months
  Assessment of the presence or absence of AMD.

SECONDARY OUTCOMES:
To evaluate how diet, physical activity level, body mass index, smoking, and chronic medication correlate with the development of AMD, determining if they are protective or risk factors. | 18 months
  To characterize the environmental and lifestyle factors that may affect or influence the development of AMD.
Genetically characterize the population and the presence of common and rare variants associated with AMD. | 18 months
  To genetically characterize the inland population of Lousã and assess the presence of common and rare variants associated with AMD.
The 10-year incidence of AMD in the inland population. | 18 months
  To determine the 10-year incidence of AMD in the inland population, and compare it and analyze together with the coastal population cohort 5-year incidence.
Identify genotypic-phenotypic correlations. | 18 months
  To establish genotypic-phenotypic correlations (both rare and common variants) in either cohort and for the total population.

CONTACTS AND LOCATIONS:
Locations (1):
- AIBILI-CEC (AIBILI- Clinical Trials Centre), Coimbra, Portugal